CLINICAL TRIAL: NCT01439802
Title: Transcesarean IUD Insertion: A Prospective Cohort Study
Brief Title: Copper Intrauterine Device (IUD) Insertion at Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2007-345-002
Record Dates: First submitted 2011-09-21; First posted 2011-09-23 (Estimated); Results first posted 2022-12-29 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Intrauterine Device Expulsion
Keywords: Postpartum IUD; Cesarean Delivery; 6 months postpartum; satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Copper IUD placement at time Cesarean Delivery (Copper T 380A) — Placement of Paragard IUD at time of Cesarean Delivery
  Other Names: Copper T 380A

SUMMARY:
The purpose of this study is to determine the expulsion rates of copper Intrauterine Devices (IUDs) placed at time of Cesarean Delivery.

DETAILED DESCRIPTION:
This was a prospective clinical study with 90 patients undergoing cesarean section. After delivery of the placenta, a ParaGard® copper T380A IUD was inserted through the hysterotomy site. IUD placement was confirmed by visualization of the strings at the cervical os or via ultrasound at the 6 week postpartum visit. Subjects also received a phone call 6 months after IUD placement to ascertain physician follow-up and patient satisfaction. This telephone call was to ensure that each subject attended her postpartum visit, had an evaluation of IUD placement and then we performed a survey. This survey used a Likert Scale to measure each subject's satisfaction. The fields included very satisfied, satisfied, somewhat satisfied, neutral, somewhat unsatisfied, unsatisfied and very unsatisfied.

ELIGIBILITY:
Inclusion Criteria:

* singleton gestation
* greater than 35 weeks gestation
* speaks English or Spanish
* desires IUD for contraception
* undergoing a cesarean delivery

Exclusion Criteria:

* evidence of chorioamnionitis
* history of chlamydia within this pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2008-08; Primary Completion 2009-11 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amitasrigowri Murthy, MD, Principal Investigator — NYU School of Medicine
Locations (2):
- United States (2):
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center, Weiler Division, The Bronx, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place in two Bronx medical centers. During prenatal care, all women were counseled regarding contraception. Women who intended to use the copper T380A IUD postpartum were approached and informed about the study after arriving on labor and delivery. Women undergoing cesarean delivery at >= 35 weeks of gestation and who met all of the inclusion and none of the exclusion criteria were enrolled into the study upon signing informed consent.
Groups:
- Postplacental Insertion of Intrauterine Device (IUD): This was a single arm study. All patients were enrolled into the Postplacental Insertion of Copper T380A IUD arm/group.
  IUDs were placed into the endometrial cavity through the uterine incision immediately after delivery of the infant and placenta. The IUD was removed from its applicator and manually placed in the most proximal part of the endometrial cavity. Ring forceps were used to place the strings into the cervix. IUD strings were not trimmed at the time of insertion.
Period: 6 Weeks Postpartum Status
Arm/Group | Postplacental Insertion of Intrauterine Device (IUD)
Started | 90
Completed | 54
Not Completed | 36
Not completed — Lost to Follow-up | 36
Period: 6 Months Postpartum Status
Arm/Group | Postplacental Insertion of Intrauterine Device (IUD)
Started | 54
Completed | 42
Not Completed | 12
Not completed — Lost to Follow-up | 12

BASELINE CHARACTERISTICS:
Arm/Group | Postplacental Insertion of Intrauterine Device (IUD)
Number analyzed (Participants) | 90
Age, Customized [Count of Participants; unit: Participants]
  <20 years old | 2
  20-29 years old | 40
  30-39 years old | 45
  40-49 years old | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 31
  Hispanic | 46
  Asian | 4
  Other | 2
  Not Specified | 7
Region of Enrollment [Number; unit: participants]
  United States | 90
Parity [Count of Participants; unit: Participants] — Nulliparous participants were identified as those who had no previous childbirths and Multiparous participants were defined as those that had at least one previous childbirth.
  Participants
    Nulliparous | 4
    Multiparous | 86
Indication [Count of Participants; unit: Participants] — Overall count of 91 participants as the indication categories were not considered to be mutually exclusive (i.e., more than 1 indication could have been selected for participants who were not categorized as 'Elective Repeat').
  In this context, indication describes the condition the participant presented with during consent and enrollment into the study.
  Participants
    Elective Repeat | 66
    Shoulder Dystocia | 5
    Macrosomia | 8
    Malpresentation | 5
    Preeclampsia | 3
    Other | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Expulsion of IUD
Description: Number of participants with Expulsion of IUDs placed at time of cesarean delivery.
Time Frame: 6 week postpartum
Population: Fifty-four (54) of ninety (90) participants were able to be reached for a response at 6 weeks either in person or via telephone.
Measure: Count of Participants; unit: Participants
Arm/Group | Postplacental Insertion of Intrauterine Device (IUD)
Number analyzed (Participants) | 54
Participants
  IUD Maintained | 54
  IUD Expelled | 0

2. Secondary Outcome: Satisfaction of IUD Placement
Description: Satisfaction of subjects who received an IUD at time of cesarean delivery was measured based on a telephone survey administered 6 months postpartum. A 4-point Likert scale ("Very Happy/Happy", "Somewhat Happy", "Unsure", "Unhappy") was used to evaluate participants' attitude toward the IUD.
Time Frame: 6 months postpartum
Population: Forty-two (42) of the ninety (90) enrolled participants were able to be reached at 6 months following IUD placement.
Measure: Count of Participants; unit: Participants
Arm/Group | Postplacental Insertion of Intrauterine Device (IUD)
Number analyzed (Participants) | 42
Participants
  Very Happy/Happy | 34
  Somewhat Happy | 4
  Unsure | 4
  Unhappy | 0

3. Secondary Outcome: Number of Participants With Expulsion of IUD
Description: Number of participants with Expulsion of IUDs placed at time of cesarean delivery.
Time Frame: 6 months postpartum
Population: Forty-two (42) of ninety (90) participants were able to reached at 6 months following IUD placement.
Measure: Count of Participants; unit: Participants
Arm/Group | Postplacental Insertion of Intrauterine Device (IUD)
Number analyzed (Participants) | 42
Participants
  IUD Maintained | 42
  IUD Expelled | 0

ADVERSE EVENTS:
Time Frame: 6 months postpartum
Arm/Group | Postplacental Insertion of Intrauterine Device (IUD)
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 23/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Postplacental Insertion of Intrauterine Device (IUD) (N=42)
Heavy menstrual bleeding (Pregnancy, puerperium and perinatal conditions) | 6 (6)
Cramping (Pregnancy, puerperium and perinatal conditions) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No